CLINICAL TRIAL: NCT06764836
Title: An Open-Label, Multi-Centre, Single-Arm, Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Antitumor Efficacy of IMM2510 in Combination With IMM27M in Patients With Advanced Solid Tumors
Brief Title: A Study of IMM2510 + IMM27M Combination Therapy in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: ImmuneOnco Biopharmaceuticals (Shanghai) Inc. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMM2510-002
Record Dates: First submitted 2024-12-22; First posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Advanced Solid Tumors; HCC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IMM2510 + IMM27M Combination Therapy (Experimental): Dose Escalation Phase:
  Participants will receive IMM27M 3.0 mg/kg single dose on day 1 (C1D1), and after a 4-week interval, will receive IMM2510 10.0 mg/kg or 20.0 mg/kg dose every 2 weeks (Q2W).
  Dose Expansion Phase:
  The dose of IMM27M and IMM2510 for the dose expansion phase is determined according to the dose escalation results.
  Participants will receive IMM27M single dose on day 1 (C1D1), and after a 4-week interval, will receive IMM2510 every 2 weeks (Q2W).
  Interventions: Drug: IMM27M; Drug: IMM2510

INTERVENTIONS:
Drug: IMM27M — Intravenous injection
Drug: IMM2510 — Intravenous injection

SUMMARY:
This study is an open-label, multi-centre, single-arm, phase I clinical study, to evaluate the safety, tolerability, efficacy, pharmacokinetics (PK) and pharmacodynamics (PD) of IMM2510 (an anti-PD-L1/VEGF bispecific antibody fusion protein) + IMM27M (a humanized Fc-engineered anti-CTLA-4 antibody) combination therapy in patients with advanced solid tumors.

DETAILED DESCRIPTION:
Dose Escalation Phase: 3+3 Dose escalation design of IMM27M + IMM2510 combination therapy in advanced solid tumors.

Dose Expansion Phase: Recommended dose for expansion (RDE) of IMM27M + IMM2510 combination therapy in three cohorts: cohort 1: locally advanced unresectable or metastatic triple-negative breast cancer (those with at least first-line systemic treatment failure or intolerance); cohort 2: advanced hepatocellular carcinoma (patients with at least first-line systemic therapy failure or intolerance); cohort 3: other advanced solid tumors (those with at least first-line systemic treatment failure or intolerance).

ELIGIBILITY:
Inclusion Criteria:

1. The patient can understand the procedures and methods of this clinical trial. After giving full informed consent, the patient voluntarily participates in it and signs the informed consent form.
2. Aged between 18 and 75 years old (including both ends), regardless of gender.
3. Clinical diagnosis:

   Dose escalation phase: Patients with advanced malignant solid tumors confirmed by histology or cytology, who have failed previous standard treatments, have no standard treatment regimens or are not suitable for standard treatment at present, including but not limited to hepatocellular carcinoma, triple-negative breast cancer, soft tissue sarcoma, non-small cell lung cancer, epithelial ovarian cancer, small cell lung cancer, malignant melanoma, colorectal cancer, ovarian cancer, endometrial cancer, renal cell carcinoma, squamous cell carcinoma of the head and neck, etc.

   Dose expansion phase: The following tumor types are included: a. Patients with advanced hepatocellular carcinoma who have failed or could not tolerate at least one line of previous systemic treatment; b. Patients with locally advanced, unresectable or metastatic triple-negative breast cancer confirmed by histology or cytology, who have failed or could not tolerate at least one line of previous systemic treatment; c. Patients with other advanced malignant solid tumors (except those with triple-negative breast cancer and advanced hepatocellular carcinoma) confirmed by histology or cytology, who have failed or could not tolerate at least one line of previous systemic treatment, including but not limited to soft tissue sarcoma, non-small cell lung cancer, epithelial ovarian cancer, small cell lung cancer, malignant melanoma, colorectal cancer, ovarian cancer, endometrial cancer, renal cell carcinoma, squamous cell carcinoma of the head and neck, etc.
4. Dose escalation phase: According to RECIST version 1.1, there should be at least one evaluable tumor lesion; Dose expansion phase: According to RECIST version 1.1, there should be at least one measurable tumor lesion.
5. ECOG performance status score of 0 - 1.
6. The expected survival time is more than 3 months.
7. There should be sufficient organ function. Hematological system (without receiving blood transfusion or hematopoietic stimulating factor treatment within 14 days): Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L, Platelet count (PLT) ≥ 100 × 10⁹/L, Hemoglobin (Hb) ≥ 90 g/L. For patients with HCC accompanied by liver cirrhosis, ANC ≥ 1.0 × 10⁹/L and platelet count ≥ 90 × 10⁹/L are acceptable for enrollment.

   Liver function: Total bilirubin (TBIL) ≤ 1.5 × upper limit of normal (ULN), for patients with liver metastasis or liver cancer, TBIL ≤ 3.0 × ULN; Alanine aminotransferase (ALT) ≤ 2.5 × ULN, for patients with liver metastasis or liver cancer, ALT ≤ 5.0 × ULN; Aspartate aminotransferase (AST) ≤ 2.5 × ULN, for patients with liver metastasis or liver cancer, AST ≤ 5.0 × ULN.

   Renal function: Creatinine clearance rate (Ccr) ≥ 50 ml/min (calculated according to the Cockcroft-Gault formula), Urinary protein < 2+ or 24-hour urinary protein quantification < 1.0 g.

   Coagulation function: Prothrombin time (PT) ≤ 1.5 × ULN, Activated partial thromboplastin time (APTT) ≤ 1.5 × ULN, International normalized ratio (INR) ≤ 1.5 × ULN.

   Cardiac function: 12-lead electrocardiogram, QTc interval ≤ 480 ms, Echocardiogram, Left ventricular ejection fraction (LVEF) ≥ 50%.

   Thyroid function: Thyroid-stimulating hormone (TSH) ≤ 1 × ULN (if abnormal, FT3 and FT4 levels should be observed simultaneously. If FT3 and FT4 levels are normal, enrollment is allowed).

   Liver function grading for HCC patients: Child-Pugh score ≤ 7 points.
8. Qualified patients (both male and female) with fertility must agree to use reliable contraceptive methods (hormonal or barrier methods or abstinence) together with their partners during the trial period and at least 6 months after the last administration.
9. The patient must be informed of this study before the trial and voluntarily sign the written informed consent form.

Exclusion Criteria:

Patients meeting any one of the following criteria will be excluded from this study:

1. Previous treatment history:

   1. Patients who received mitomycin and nitrosourea chemotherapy within 6 weeks before the first administration.
   2. Patients who received the last systemic anti-tumor treatment, including chemotherapy, radiotherapy, immunotherapy, biological agents or endocrine therapy, etc., within 4 weeks before the first administration.
   3. Patients who received hormonal anti-tumor treatment or small molecule targeted therapy within 2 weeks before the first administration.
   4. Patients who received local treatment such as radiotherapy for target lesions within 4 weeks before the first administration, and those who received palliative local treatment for non-target lesions within 2 weeks before the first administration.
   5. Patients who received non-specific immunomodulatory treatment (such as interleukin, interferon, thymosin, tumor necrosis factor, etc., excluding IL-11 used for treating thrombocytopenia) within 2 weeks before the first administration.
   6. Patients who previously received the experimental drugs IMM2510 and/or IMM27M; those who could not tolerate treatment with anti-CTLA-4 or PD-1/L1 inhibitors (due to toxic and side effects); those who previously used drugs targeting three targets, namely anti-PD-1/L1, VEGF, and CTLA-4 simultaneously in the same regimen.
   7. Patients who received traditional Chinese medicine with anti-tumor indications within 1 week before the first administration.
   8. Patients who participated in other clinical trials within 4 weeks before the first administration.
2. Those with a known severe allergic history to any component of the experimental drug, or those with a history of severe allergic reactions to chimeric or humanized antibodies or fusion proteins.
3. Those who had any immune-related adverse events (irAE) of grade ≥ 3 in CTCAE V5.0 or that led to the termination of immunotherapy during previous treatment with any immunotherapy drugs.
4. Those diagnosed with other malignant tumors within 5 years before enrollment. Exceptions: 1) Cervical carcinoma in situ and non-melanoma skin cancer that have been cured; 2) Patients who have been radically cured, unless the patients have been in complete remission for at least 2 years before enrollment and do not require other treatments or will not require other treatments during the study period.
5. Those with an active second primary cancer that is known and has had no recurrence within 5 years. Exceptions: 1) The investigator believes that both primary cancers can benefit from this study; 2) The investigator has clearly excluded which primary tumor the metastatic lesions belong to.
6. Patients with primary central nervous system (CNS) malignant tumors or those with active CNS metastases that failed local treatment (radiotherapy or surgical treatment). However, the following patients are allowed to enroll: a. Patients with asymptomatic brain metastases; b. Patients with clinically stable symptoms (i.e., no radiological progression was seen within 4 weeks before the first administration, and any neurological symptoms have returned to the baseline level), and who have not required corticosteroid hormones and other treatments for brain metastases for ≥ 4 weeks.
7. Patients with hypertension that cannot be controlled by drugs (systolic blood pressure remains > 140 mmHg or diastolic blood pressure > 90 mmHg after standard treatment), or with pulmonary hypertension or unstable angina pectoris; those who had a myocardial infarction or underwent bypass or stent surgery within 6 months before administration; those with a history of chronic heart failure of grade 3 - 4 according to the New York Heart Association (NYHA) criteria; those with clinically significant valvular diseases; those with severe arrhythmias requiring treatment (except atrial fibrillation and paroxysmal supraventricular tachycardia), including QTcF ≥ 450 ms for men and ≥ 470 ms for women (calculated by the Fridericia formula); those with cerebrovascular accidents (CVA) or transient ischemic attacks (TIA), etc., within 12 months before enrollment.
8. Those with a history of arterial thrombosis, deep vein thrombosis or pulmonary embolism within 3 months before administration.
9. Those with a history of moderate or severe dyspnea at rest due to advanced malignant tumors or their complications or severe primary lung diseases, or those currently requiring continuous oxygen inhalation treatment, or those with a history of interstitial lung disease (ILD) or pneumonia, severe chronic obstructive pulmonary disease, severe pulmonary insufficiency, symptomatic bronchospasm, etc.
10. Those with diseases that may cause gastrointestinal bleeding or perforation (such as duodenal ulcer, intestinal obstruction, acute Crohn's disease, ulcerative colitis, extensive resection of the stomach and small intestine, etc.); patients with chronic Crohn's disease and ulcerative colitis (except those who have undergone total colectomy and rectal resection) should be excluded even during the inactive period; those with hereditary non-polyposis colorectal cancer or familial adenomatous polyposis syndrome; those with a history of intestinal perforation or intestinal fistula that have not been cured after surgical treatment; esophageal and gastric varices; or the presence of cancer thrombus in the main portal vein; those requiring repeated drainage due to uncontrollable thoracic, abdominal or pericardial effusion that requires puncture and drainage treatment or those with obvious symptoms.
11. Those with evidence of severe active infections that cannot be controlled (such as sepsis, bacteremia, viremia, etc.).
12. Those with active tuberculosis infection.
13. Those with active hepatitis B (HBsAg positive, and HBV DNA higher than the lower limit of detection, and excluding hepatitis caused by drugs or other reasons), or those with active hepatitis C (anti-HCV antibody positive, and HCV RNA higher than the lower limit of detection).
14. Those with a history of immunodeficiency, including human immunodeficiency virus (HIV) infection, or other immunodeficiency diseases, or those with a history of organ transplantation or hematopoietic stem cell transplantation.
15. Those with a history of active autoimmune diseases, including but not limited to systemic lupus erythematosus, psoriasis, rheumatoid arthritis, inflammatory bowel diseases, Hashimoto's thyroiditis, autoimmune thyroid diseases, multiple sclerosis, etc. Exceptions:

    1. Hypothyroidism that can be controlled only by hormone replacement therapy.
    2. Skin diseases that do not require systemic treatment (such as vitiligo, psoriasis).
    3. Controlled celiac disease.
16. Those who are currently using immunosuppressants or systemic hormone therapy (prednisone at a dose of ≥ 10 mg/day or other equivalent hormones) and are still using them within 2 weeks before enrollment.
17. Those who underwent major surgery within 4 weeks before the first administration and have not fully recovered, or those who plan to undergo major surgery within the first 12 weeks after receiving the study drug; those who received minor surgical operations 2 days before enrollment.
18. Those with incompletely healed skin wounds, surgical sites, trauma sites, severe mucosal ulcers or fractures, and whom the investigator judges to be at risk of bleeding if participating in this study.
19. Those who received anti-tumor vaccines or live vaccines within 4 weeks before the first administration, or those who plan to receive anti-tumor vaccines or live vaccines during the study period.
20. Those with a clear history of neurological or mental disorders in the past, such as epilepsy, dementia, and with poor compliance.
21. Patients with a history of alcoholism or drug abuse within the past year, or with a history of fainting during acupuncture or blood drawing, or those who cannot tolerate venipuncture for blood collection.
22. Women who are pregnant or breastfeeding; those who do not agree to take sufficient contraceptive measures together with their partners during the study period and within 6 months after the end of receiving the experimental drug.
23. The investigator believes that there are other reasons why the patient is not suitable to participate in this trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2026-01-27 (Estimated); Study Completion 2026-01-27 (Estimated)

PRIMARY OUTCOMES:
DLT/MTD (Dose Escalation Phase) | Within 8 weeks after the investigational products administration (within 56 days after first dosing of C1D1)
  Incidence and characteristics of Dose-Limiting Toxicity (DLT) to determine the Maximum Tolerated Dose (MTD).
RP2D (Dose Extension Phase) | From the first dose until disease progresses or end of treatment for other reasons, the maximum treatment duration is not more than 48 weeks
  Recommended Phase II Dose (RP2D) of IMM27M and IMM2510, as the dose for efficacy study in Phase II, will be the dose with promising clinical responses observed in the patients, and well tolerated by patients.
Incidence and characteristics of AEs and SAEs (according to NCI CTCAE 5.0) | From the first dose to 30 days after the last dose [90 days for SAEs and Immune-related Adverse Event (irAEs) ], or until beginning new anti-tumor treatment
  Incidence and characteristics of Adverse Events (AEs) and Serious Adverse Events (SAEs) throughout the study period, were evaluated according to Common Terminology Criteria for Adverse Events (CTCAE) V5.0.

SECONDARY OUTCOMES:
ORR | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years
  Objective Response Rate (ORR) is the proportion of patients with Complete Response (CR) or Partial Response (PR). ORR and other efficacy evaluation indexes are based on RECIST 1.1 criteria, the iRECIST criteria is supplemental only.
DCR | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years
  Disease control rate (DCR) is the proportion of patients with CR, PR, and Stable Disease (SD).
DOR | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years
  Duration of Response (DOR) is the time between the first onset of CR or PR and the first onset of Disease Progression (PD) or death from any cause. For patients with unknown progression or death, the time of sustained remission was censored at the time point of the last patient evaluation.
PFS | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years
  Progression-Free Survival (PFS) is the time between first initiation of study treatment to PD or death due to any reason. For patients with unknown progression or death, disease-free survival was censored at the time point of the last patient evaluation.
OS | From date of first dose until the date of first documented progression, death from any cause, loss of follow-up, withdrawal of informed consent, or study termination by the sponsor, whichever came first, assessed up to approximately 2 years
  Overall Survival (OS) is defined as the time interval from the date of the first dose of study drug to the date of death from any cause.
Cmax | Up to approximately 1 year
  Peak concentration (Cmax), in single dose period.
Tmax | Up to approximately 1 year
  Peak time (Tmax), in single dose period.
t1/2 | Up to approximately 1 year
  Elimination phase half-life (t1/2), in single dose period.
AUC0-t | Up to approximately 1 year
  Area under plasma concentration-time curve from 0 to the last quantifiable time point (AUC0-t), in single dose period.
AUC0-∞ | Up to approximately 1 year
  Area under plasma concentration-time curve from 0 to infinite time (AUC0-∞), in single dose period.
Cmin, ss | Up to approximately 1 year
  Steady-state trough concentration (Cmin, ss), in multiple dose periods.
Cmax, ss | Up to approximately 1 year
  Steady-state peak concentration (Cmax, ss), in multiple dose periods.
Tmax, ss | Up to approximately 1 year
  Steady-state peak time (Tmax, ss), in multiple dose periods.
t1/2, ss | Up to approximately 1 year
  Steady-state half-life (t1/2, ss), in multiple dose periods.
Cav, ss | Up to approximately 1 year
  Mean plasma concentration at steady state (Cav, ss), in multiple dose periods.
ADA and NAb | Up to approximately 1 year
  For each patient, the presence of Anti-drug Antibody (ADA) will be assessed, and ADA positive patients need to be measured for titers and Neutralizing Antibodies (NAb).

CONTACTS AND LOCATIONS:
Locations (1):
- ZhongShan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No